CLINICAL TRIAL: NCT02116231
Title: Phase II Study Comparing Intensity Modulated Radiotherapy (IMRT) in Combination With Concurrent Chemotherapy and IMRT Alone for Stage II Nasopharyngeal Carcinoma
Brief Title: The Role of Adding Concurrent Chemotherapy to IMRT in the Treatment of Stage II Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHGX20140402
Record Dates: First submitted 2014-04-02; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Effects of Chemotherapy
Keywords: Nasopharyngeal neoplasm;IMRT; Concurrent chemotherapy
MeSH Terms: interventions — Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent chemoradiotherapy (Experimental): Concurrent chemoradiotherapy: IMRT was given to the patients with regimen of 66Gy-76Gy to the gross target volume of nasopharynx,66-70Gy to the gross target volume of positive nodes, 60-62Gy the high risk clinical target volume, 50-56Gy to the low risk clinical target volume. Concurrent chemotherapy is administrated with cisplatin 100mg/m2 at d1, d22, d43 during radiotherapy.
  Interventions: Drug: Concurrent chemotherapy with cisplatin; Radiation: Intensity modulated radiotherapy
- IMRT alone (Active Comparator): IMRT is given to the patients with regimen of 66Gy-76Gy to the gross target volume of nasopharynx,66-70Gy to the gross target volume of positive nodes, 60-62Gy the high risk clinical target volume, 50-56Gy to the low risk clinical target volume.
  Interventions: Radiation: Intensity modulated radiotherapy

INTERVENTIONS:
Drug: Concurrent chemotherapy with cisplatin — Three cycles of weekly Cisplatin 100 mg/m2 starting on the first day of IMRT
  Arms: Concurrent chemoradiotherapy
Radiation: Intensity modulated radiotherapy — Intensity modulated radiotherapy is a technique of radiotherapy.

SUMMARY:
The study is designed to compare Intensity Modulated Radiotherapy (IMRT) in combination with concurrent chemotherapy and IMRT alone in treatment of stage II nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is endemic in Southern China, Southeast Asia, the Arctic, and mid-East/North Africa. NPC prevalence is reported to be highest in southern China, where an average of 80 cases per 100,000 population are reported each year. It is both radiosensitive and chemosensitive. The National Comprehensive Cancer Network (NCCN) guidelines (version 1, 2013), have recommended use of concurrent chemoradiotherapy (CCRT) with or without adjuvant chemotherapy (AC) as standard treatment for NPC.

Recently, the technique of IMRT has become widely used in the treatment of nasopharyngeal carcinoma. The preliminary results showed that IMRT might improve the rate of local control and the quality of life in NPC. In a retrospective study (Ivan,2010), the result showed that IMRT without concurrent chemotherapy provides good outcome for patients with stage IIB NPC with acceptable toxicity. Another study showed that Comparing with IMRT alone, IMRT in combination with chemotherapy provided no significant benefit to locoregionally advanced NPC (Su,2011). With IMRT, it was unclear whether the additional of concurrent chemotherapy was essential for stage II nasopharyngeal carcinoma.

The investigators designed the present study to research the role of adding concurrent chemotherapy to intensity modulated radiotherapy in the treatment of stage II NPC. The primary endpoint is failure-free survival (FFS).The second endpoints were overall survival (OS),loco-regional failure-free survival (LFFS), distant metastasis failure-free survival (DMFS), and acute and late adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type).
* 18 Years to 70 Years
* Tumor staged as T1-2N1/ T2N0 (according to the 7th AJCC edition),No evidence of distant metastasis (M0)
* Satisfactory performance status: Karnofsky scale (KPS) > 70 (Appendix I ).
* Adequate marrow: leucocyte count > 4×109/L, neutrophil count > 2×109/L, hemoglobin > 90g/L and platelet count > 100×109/L
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) < 2.5×ULN, and bilirubin < ULN
* Adequate renal function: creatinine clearance > 60 ml/min
* Patients must be informed of the investigational nature of this study and give written informed consent

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Age > 60 or < 18.
* Treatment with palliative intent.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | One year
  The time is calculated from the date of diagnosis to the date of occurrence of relapse or distant metastasis.

SECONDARY OUTCOMES:
Overall survival (OS) | One year
  The time is calculated from the date of diagnosis to the date of patient death.
Loco-regional failure-free survival (LFFS) | One year
  The time is calculated from the date of diagnosis to the date of a relapse of local or nodal tumors.
Distant metastasis failure-free survival (DMFS) | One year
  The time is calculated from the date of diagnosis to the date of occurrence of relapse or distant metastasis.
Acute and late adverse events | Four months
  The side effects will be evaluated according to CTCAE V 3.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Guangxi Medical University, Nanning, Guangxi, China

REFERENCES:
- [Background] Yoshizaki T, Ito M, Murono S, Wakisaka N, Kondo S, Endo K. Current understanding and management of nasopharyngeal carcinoma. Auris Nasus Larynx. 2012 Apr;39(2):137-44. doi: 10.1016/j.anl.2011.02.012. Epub 2011 May 17. PMID 21592702
- [Background] Chan AT, Teo PM, Johnson PJ. Nasopharyngeal carcinoma. Ann Oncol. 2002 Jul;13(7):1007-15. doi: 10.1093/annonc/mdf179. PMID 12176778
- [Background] Su SF, Han F, Zhao C, Huang Y, Chen CY, Xiao WW, Li JX, Lu TX. Treatment outcomes for different subgroups of nasopharyngeal carcinoma patients treated with intensity-modulated radiation therapy. Chin J Cancer. 2011 Aug;30(8):565-73. doi: 10.5732/cjc.010.10547. PMID 21801605
- [Background] Tham IW, Lin S, Pan J, Han L, Lu JJ, Wee J. Intensity-modulated radiation therapy without concurrent chemotherapy for stage IIb nasopharyngeal cancer. Am J Clin Oncol. 2010 Jun;33(3):294-9. doi: 10.1097/COC.0b013e3181d2edab. PMID 20395788
- See also: Guangxi Medical University — http://www.gxmu.edu.cn/